CLINICAL TRIAL: NCT06219070
Title: Effect of Core Training on Physical Fitness and Smash Performance Among Female Badminton Players in Guangxi, China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ma Shuzhen (Other)
Responsible Party: Sponsor-Investigator, Ma Shuzhen, lecturership, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Ma Shuzhen
Record Dates: First submitted 2024-01-07; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Athletes
Keywords: Core training; Physical fitness; Smash performance; Female badminton Players

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Their information may need to be kept confidential
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will undergo 60 minutes of Core Training.
  Interventions: Other: Core straining
- Control group (No Intervention): The control group will follow the curriculum standards set by the Sports University.

INTERVENTIONS:
Other: Core straining — The experimental group received 12 weeks of core training, and the control group received 12 weeks of conventional training, 3 times/times Of the week. Each session lasts 60 minutes and includes warm-up, exercise, and relaxation.
  Arms: Experimental group

SUMMARY:
The performance of Chinese women's badminton singles players is declining to a large extent, the training of badminton in China needs to catch up, and the talent ladder has caused a fault. Badminton Routine training, the effect is not apparent . An essay on the impact of core training on athletes' skill performance was written by Luo; it proves that core strength training plays a positive role in a variety of sports; there is no study of female badminton players. Coaches or sports researchers can use this knowledge to manage the training load of badminton players better, thereby helping badminton players achieve better results in badminton training and competition.

DETAILED DESCRIPTION:
Hibbs constructed the Model of Core Training and Potential Performance according to the theoretical framework of core strength training. This study intervention design part of the researchers referred to Greg Glassman's "CrossFit training guide" and theoretical framework of core strength training. Motion design source form Motion design source "Diversified Training to Enhance Core Strength State General Administration of sport (Sport.gov.cn)"and Khatoon wrote the article. The duration and frequency of intervention came from the review. It is found in reviewing the effect of core strength training on badminton players' performance is 8 weeks and 3 times. Therefore, this study adopted intervention for 8 weeks, 3 times a week. The subjects of this study are 18-22 years old female college elite badminton players, all of whom are national second-level and above athletes. This study employs a Cluster Randomized Controlled Trial (CRCT) design. The athletes were randomly assigned to two training sites and divided into experimental and control groups. The two groups had the same professional skills training content. The only difference was the physical training part. The training program of the two groups lasts 8 weeks, 3 times per week, and 1 hour per training. The experimental group performed core training, while the control group maintained routine training. In addition, the specific content of the routine training of the control group was the standard training plan of the school. The dependent variables measured in this study are physical fitness (strength, speed, endurance, agility, and flexibility) and killing the ball under different states, including in sit Smash, jump smash, move left smash, move right smash, and back smash.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-22 years.
2. Chinese university female badminton players.
3. No sports injuries, such as ankle injuries or waist injuries.
4. Elite athlete

Exclusion Criteria:

1. Athletes who were systematically training their core strength.
2. Athletes with sports injuries such as ankle or waist injuries.
3. Who could not follow the entire training schedule for three months.
4. Students who work out regularly or have hobbies for extra physical exercise.
5. Students with physical or mental illness.

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2024-05-05 (Estimated); Study Completion 2024-08-05 (Estimated)

PRIMARY OUTCOMES:
Effects of strength among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  Measure the distance of the standing long jump with a measuring tape in centimeters (cm).
Effects of endurance among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  Recorded the number of jumping ropes in 1 min.
Effects of Speed among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  Use a stopwatch to record the time taken by the athlete to run 20 times with a low center of gravity (measured in seconds)
Effects of agility among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  The course measured 10 meters in length and 5 meters in width when it was set up on a basketball court. The start, finish line, and both turning points were indicated by four cones. Four more cones were positioned at equal intervals down the center. The distance between the central cones was 3.3 meters. To cross the finish line, the subjects were told to run as fast as they could around the course in the designated direction. Time spent recording (seconds)
Effects of flexibility among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  Use the sit-and-reach box. The score is recorded as the point where their fingertips reach the measurement scale. The range of motion is measured in cm.
Effects of In sit Smash among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  Accuracy and velocity test
Effects of Jump smash among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  The athlete's task was to perform such a shot that the shuttlecock flew between the net and the colored string, giving the shuttlecock the highest possible velocity, Badminton subjects use their own rackets (according to the player's personal preferences) to spike the ball, test 10 balls, and record the number successful of 10 balls(times), and use a SMART BDMINTON SENSOR to record the speed of each ball（km/h）. The test process is as follows in sit smash, jump smash, move left smash, move right smash, back smash.
Effects of move left smash among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  The athlete's task was to perform such a shot that the shuttlecock flew between the net and the colored string, giving the shuttlecock the highest possible velocity, Badminton subjects use their own rackets (according to the player's personal preferences) to spike the ball, test 10 balls, and record the number successful of 10 balls(times), and use a SMART BDMINTON SENSOR to record the speed of each ball（km/h）. The test process is as follows in sit smash, jump smash, move left smash, move right smash, back smash.
Effects of move right smash among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  The athlete's task was to perform such a shot that the shuttlecock flew between the net and the colored string, giving the shuttlecock the highest possible velocity, Badminton subjects use their own rackets (according to the player's personal preferences) to spike the ball, test 10 balls, and record the number successful of 10 balls(times), and use a SMART BDMINTON SENSOR to record the speed of each ball（km/h）. The test process is as follows in sit smash, jump smash, move left smash, move right smash, back smash.
Effects of back smash among college students | Pretest : before intervention Post-test 1 : 4 weeks after intervention Post-test 2 : 8 weeks after intervention
  The athlete's task was to perform such a shot that the shuttlecock flew between the net and the colored string, giving the shuttlecock the highest possible velocity, Badminton subjects use their own rackets (according to the player's personal preferences) to spike the ball, test 10 balls, and record the number successful of 10 balls(times), and use a SMART BDMINTON SENSOR to record the speed of each ball（km/h）. The test process is as follows in sit smash, jump smash, move left smash, move right smash, back smash.

CONTACTS AND LOCATIONS:
Overall Officials: kims@upm.edu.my Soh, Study Director — Universiti Putra Malaysia
Locations (1):
- Ma Shuzhen, Guangxi, China

IPD SHARING:
Plan to Share IPD: No